CLINICAL TRIAL: NCT01049529
Title: Efecto Modulador de la Administracion Del Acido Docosahexaenoico Sobre la Respuesta Inflamatoria, la evolución Clinica y el Estado Nutricional de Neonatos Sometidos a cirugía
Brief Title: Effect of Docosahexaenoic Acid on the Inflammatory Response and Clinical Outcomes From Surgical Patients
Acronym: DHA-IRCO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Mariela Bernabe García, Researcher, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2005/3603/72; 2005/1/I/193 (Other Grant/Funding Number: Fondo para la Investigación en Salud, IMSS)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Severe Sepsis; Organ Dysfunction Syndrome
Keywords: Docosahexaenoic acid; n-3 Long Chain Polyunsaturated Fatty Acids; omega 3 fatty acids; neonates; clinical outcomes; critically ill patients; Inflammatory and antiinflammatory cytokines; Length of intensive care stay
MeSH Terms: conditions — Sepsis | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (Placebo Comparator): This group is receiving sunflower oil (the excipient for DHA)
  Interventions: Dietary Supplement: Placebo
- DHA group (Active Comparator): This group is receiving the docosahexaenoic acid (DHA) supplement
  Interventions: Dietary Supplement: Docosahexaenoic acid

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid — DHA have oil form. Each neonate is receiving 75 mg/kg/day of DHA in 188 uL/kg/day in two doses per day, since two days before surgery and over six days following cardiovascular surgery
  Other Names: n-3 LC-PUFAs; omega 3 fatty acids; Long chain polyunsaturated fatty acids
  Arms: DHA group
Dietary Supplement: Placebo — Placebo have oil form. Each neonate is receiving 188uL/kg/day of sunflower oil as placebo in two doses per day, since two days before surgery and over six days following cardiovascular surgery
  Other Names: Life's DHA
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate if enteral docosahexaenoic acid (DHA) administration attenuates the inflammatory cytokines and improve clinical outcomes in neonates who underwent cardiovascular surgery

DETAILED DESCRIPTION:
Severe sepsis and organ failure are leading causes of death in surgical patients. Several studies indicate that a causal relationship exists between the surgical or traumatic injury and the predisposition to develop septic/infectious complications and multiple organ failure; this is attributable to uncontrolled inflammatory response. Since neonates have an immature immune system, they are in a higher risk to develop uncontrolled inflammatory response and adverse clinical outcomes.

N-3 long chain polyunsaturated fatty acids (L-PUFAs) such as docosapentaenoic and docosahexaenoic acids (EPA and DHA) have been shown to reduce the inflammatory response by reducing cytokines, infection rates and length of hospitalization in patients with abdominal surgery. Therefore, acute and enteral administration of DHA may improve clinical outcomes in neonates with cardiovascular surgery

ELIGIBILITY:
Inclusion Criteria:

* Authorization from both parents for recruiting of the neonate into the study with consent signed form after the purpose and procedures have been explained
* Gestational age older than 32 weeks
* Adequate weight for gestational age
* Gastrointestinal tract that allows tolerate the doses of DHA or placebo
* No signs of Systemic Inflammatory Response Syndrome before the surgery as fever >38 degrees C or hypothermia <36 degrees C, or leukocytosis >19,500 cells/cubic mm or < 5000 cells/cubic mm or > 10% immature forms.

Exclusion Criteria:

* Fasting for more than two days after surgery
* Discharge to other hospital outside the metropolitan area
* Parents who decide to decline of the study
* Patients who necessitate cardiovascular bypass

Ages: 1 Day to 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2007-03; Primary Completion 2011-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Inflammatory response measured by cytokines IL-1, IL-6, TNF-alfa, IL-10 e IL-1ra and clinical outcomes assessed as frequency of severe sepsis, respiratory and cardiovascular dysfunction. | During the hospital stay, two weeks in average

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Bernabe-Garcia, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unit of Research in Nutrition, Pediatric Hospital, Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Alarcon M, Bernabe-Garcia M, Del Prado M, Rivera D, Ruiz G, Maldonado J, Villegas R. Docosahexaenoic acid administered in the acute phase protects the nutritional status of septic neonates. Nutrition. 2006 Jul-Aug;22(7-8):731-7. doi: 10.1016/j.nut.2006.04.002. Epub 2006 Jun 5. PMID 16750345
- [Background] Lopez-Alarcon M, Bernabe-Garcia M, del Valle O, Gonzalez-Moreno G, Martinez-Basilea A, Villegas R. Oral administration of docosahexaenoic acid attenuates interleukin-1beta response and clinical course of septic neonates. Nutrition. 2012 Apr;28(4):384-90. doi: 10.1016/j.nut.2011.07.016. Epub 2011 Nov 12. PMID 22079797
- [Result] Bernabe-Garcia M, Lopez-Alarcon M, Villegas-Silva R, Mancilla-Ramirez J, Rodriguez-Cruz M, Maldonado-Hernandez J, Chavez-Rueda KA, Blanco-Favela F, Espinoza-Garcia L, Lagunes-Salazar S. Beneficial Effects of Enteral Docosahexaenoic Acid on the Markers of Inflammation and Clinical Outcomes of Neonates Undergoing Cardiovascular Surgery: An Intervention Study. Ann Nutr Metab. 2016;69(1):15-23. doi: 10.1159/000447498. Epub 2016 Jul 9. PMID 27394149
- [Result] Bernabe-Garcia M, Lopez-Alarcon M, Salgado-Sosa A, Villegas-Silva R, Maldonado-Hernandez J, Rodriguez-Cruz M, Rivas-Ruiz R, Chavez-Sanchez L, Blanco-Favela FA, Mancilla-Ramirez J, Gordillo-Alvarez V, Madrigal-Muniz O. Enteral Docosahexaenoic Acid Reduces Analgesic Administration in Neonates Undergoing Cardiovascular Surgery. Ann Nutr Metab. 2016;69(2):150-160. doi: 10.1159/000452227. Epub 2016 Nov 2. PMID 27806350